CLINICAL TRIAL: NCT00015964
Title: A Phase II Stdy of ZD 1839 in Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: ZD 1839 in Treating Patients With Metastatic or Recurrent Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10869A; UCCRC-10869; NCI-1721
Record Dates: First submitted 2001-05-06; First posted 2004-02-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily administration of ZD1839 (Experimental)
  Interventions: Drug: ZD1839

INTERVENTIONS:
Drug: ZD1839
  Other Names: gefitinib, Iressa ®

SUMMARY:
RATIONALE: Biological therapies such as ZD 1839 may interfere with the growth of tumor cells and slow the growth of head and neck cancer.

PURPOSE: Phase II trial to study the effectiveness of ZD1839 in treating patients who have metastatic or recurrent cancer of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of ZD 1839 in patients with metastatic or recurrent squamous cell carcinoma of the head and neck. II. Determine the effectiveness of this regimen in these patients. III. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive oral ZD 1839 once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or recurrent squamous cell carcinoma of the head and neck that is incurable by surgery or radiotherapy At least 1 lesion measurable in at least 1 dimension At least 20 mm by conventional techniques OR At least 10 mm by CT scan No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 60-100% Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST/ALT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No symptomatic congestive heart failure No unstable angina pectoris No cardiac arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of allergic reactions to compounds of similar chemical or biological composition to ZD 1839 No active infection No other uncontrolled illness No psychiatric illness or social situation that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior epidermal growth factor receptor-based therapy for recurrent disease Chemotherapy: No more than 1 prior adjuvant or neoadjuvant chemotherapy and/or chemoradiotherapy regimen At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics See Chemotherapy At least 4 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics Other: No more than 1 prior regimen for recurrent disease No other concurrent investigational agents No concurrent combination antiretroviral therapy for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-03; Primary Completion 2001-09 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Early response rates of ZD1839 in head and neck tumors | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Study Chair — University of Chicago
Locations (11):
- United States (11):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Columbia LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan